CLINICAL TRIAL: NCT06359704
Title: Integrative Therapeutic Program to Regulate Expressed Emotions Among Informal Caregivers of People With Dementia: a Pilot Randomized Controlled Trial: a Study Protocol
Brief Title: Intervention for Emotions in Caregivers of Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shuangzhou Chen, Post doctoral fellow/Principal Investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: kevinszc
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: BPSD; Expressed Emotion; Depressive Symptoms
Keywords: Dementia care; Caregiver burden; Integrative intervention
MeSH Terms: conditions — Depression; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: controlled arm with waitlist treatment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPE program (Experimental): a 6-week Caregivers Of dementia Processing Emotions (COPE) program using the integrative therapy to reduce EE (primary outcome) in family caregiver of PLwD to alleviate the caregivers' depression, improve social dynamic with the PLwD, and mitigate the perceived stress from BPSD (secondary outcomes)
  Interventions: Behavioral: Caregivers Of dementia Processing Emotions (COPE) program
- Waitlist control (No Intervention): Participants in the waitlist control group, in comparison to those in the intervention group who receive treatment immediately, are placed on a waiting list and receive the same set of intervention sessions after the formal trial. This approach ensures participants have equal opportunity to receive treatment while strengthening the study's validity and overall quality by maximally controlling for potential confounding variables and biases

INTERVENTIONS:
Behavioral: Caregivers Of dementia Processing Emotions (COPE) program — a dual-modal (face-to-face and online approaches), client-customized Caregivers Of dementia Processing Emotions (COPE) program
  Arms: COPE program

SUMMARY:
This study aims to evaluate the effectiveness of a 6-week Caregivers Of dementia Processing Emotions (COPE) program using the integrative therapy to reduce EE (primary outcome) in family caregiver of PLwD to alleviate the caregivers' depression, improve social dynamic with the PLwD, and mitigate the perceived stress from BPSD (secondary outcomes).

DETAILED DESCRIPTION:
A dual-modal (face-to-face and online approaches), client-customized Caregivers Of dementia Processing Emotions (COPE) program can be developed to address EE in caregivers, such as (1) reduce caregivers' EE, (2) reduce caregivers' depressive symptoms, (3) reduce the behaviorally interactive social dynamic of maladaptation (i.e., dysfunctional dyadic relationship and quality of care), and (4) improve caregivers' perceived stress from PLwD's BPSD.

ELIGIBILITY:
Inclusion Criteria:

* with a high level of expressed emotion as indicated by a cut-off score of 35 or above on the Family Attitude Scale (Chinese version; FAS-C);(Kavanagh et al., 1997; Van Humbeeck et al., 2002; Yu et al., 2016)
* provides care at least 4 hours per day;(Moon & Adams, 2013)
* consent to participate, and
* no acute psychiatric illness.

Exclusion Criteria:

* with a low level (scored lower than 35 on FAS-C) of expressed emotion
* do not provide consistent or sufficient care (fewer than 4 hours per day) to PLwD
* do not consent to participate;
* with comorbid acute psychiatric illness.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Expressed emotions | From baseline to 3rd month followup
  Family Attitude Scale - Chinese version (FAS-C) will measure caregivers' EE (i.e., criticism and hostility) held towards the PLwD. FAS-C items are rated on a 5-point Likert scale, with higher scores indicating a higher level of EE.(Kavanagh et al., 1997; Van Humbeeck et al., 2002) Its Cronbach's alpha has been reported as 0.95, with evidence of good construct validity

SECONDARY OUTCOMES:
depressive symptoms | From baseline to 3rd month followup
  The 20-item The Centre for Epidemiologic Studies Depression (CES-D) will assess caregivers' depression, with higher scores representing greater depressive levels on a 4-point scale.(Radloff, 1977) Its internal consistency Cronbach's alpha is 0.88 in the Chinese population, while its internal reliability is 0.91 and with evidence of construct validity.(Sebern & Whitlatch, 2007; Y. Zhang et al., 2015)
social dynamics | From baseline to 3rd month followup
  Social dynamics will be measured in the aspects of dyadic relationships and quality of care. First, the 11-item Dyadic Relationship Scale (DRS) will evaluate caregivers' perspective of dyadic and family relationships in their daily caregiving activities, with a higher score indicating positive dyadic interactions; and Cronbach's alpha of 0.89 with desirable construct validity and concurrent validity.(Sebern & Whitlatch, 2007) Second, the 4-item Interaction Quality Scale (IQS) will measure the quality of care on a 6-point Likert scale, with a higher score indicating better quality of care.(Cundiff et al., 2016) IQS has desirable test-retest reliability (Cronbach's alpha = 0.96) and construct validity.(Joseph et al., 2014)
BPSD | From baseline to 3rd month followup
  The 12-item Neuropsychiatric Inventory (NPI) will assess the severity of BPSD manifested in PLwD reported by their caregivers.(Cummings, 1997) NPI comprises three levels, with higher scores indicating severer BPSD symptoms. Its test-retest reliability was 0.79 for the overall scale, and between 0.89 and 0.93 for subdomains.(Chen et al., 2018; Cummings, 1997)

CONTACTS AND LOCATIONS:
Overall Officials: Shuangzhou Chen, PhD, Principal Investigator — The University of Hong Kong